CLINICAL TRIAL: NCT07318246
Title: The Influence of Task-Oriented Learning on College Students' Creative Self-Efficacy
Brief Title: Team Work and Creative Self-Efficacy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Central Taiwan University of Science and Technology (Other)
Responsible Party: Principal Investigator, Chiu Shu-Ching, assistant professor, Central Taiwan University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2510300001
Record Dates: First submitted 2025-12-02; First posted 2026-01-05 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Self-Efficacy
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): robot backend design and control training
  Interventions: Behavioral: robot training
- control group (Other): Traditional class (not-robot )
  Interventions: Other: control group

INTERVENTIONS:
Behavioral: robot training — robot backend design and control training
  Arms: experimental group
Other: control group — Traditional class (not-robot )
  Arms: control group

SUMMARY:
This study aimed to evaluate the effects of teamwork-based task learning on college students' cognition, attitudes, skills, and creative self-efficacy, and to explore its impact within innovative technology learning contexts.

ELIGIBILITY:
Inclusion Criteria:

* Age: College students aged 18 years or older

Exclusion Criteria:

* Students who are 65 years or older, not enrolled in nursing programs, or currently on leave of absence.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Creative Self-Efficacy scale | A pre- and post-test/ up to 10 weeks
  Higher scores indicate more positive outcomes
team work scale | A pre- and post-test/ up to 10 weeks
  Higher scores indicate more positive outcomes
perception of robots | A pre- and post-test/ up to 10 weeks
  Higher scores indicate more positive outcomes
functional safety scale | A pre- and post-test/ up to 10 weeks
  Higher scores indicate more positive outcomes

SECONDARY OUTCOMES:
Reflective Journal | post-test/immediately after the intervention
  Based on your personal experience, please describe the current functions of robots or other smart technologies, your expectations for their future use in work settings, and your learning experiences with other smart technologies.

OTHER OUTCOMES:
age | Day 1
  18-65 years
sex | Day 1
  man, female
grade | Day 1
  grade1-grade 4
work1 | Day 1
  years
work2 | Day 1
  Type of job
work3 | Day 1
  Job title

CONTACTS AND LOCATIONS:
Overall Officials: Shu Ching Chiu, Principal Investigator — Central Taiwan University of Science and Technology
Locations (1):
- Central Taiwan University of Science and Technology, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No